CLINICAL TRIAL: NCT02650349
Title: StruCtuRal And FuncTional Brain Alterations by Conventional Spinal Cord Stimulation And High DensitY Stimulation: a Combined Voxel-based Morphometry and Resting State Functional Connectivity Study
Brief Title: StruCtuRal And FuncTional Brain Alterations by Conventional Spinal Cord Stimulation And High DensitY Stimulation
Acronym: SCRATCHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Moens Maarten, Prof dr., Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRATCHY1
Record Dates: First submitted 2015-12-24; First posted 2016-01-08 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Failed Back Surgery Syndrome
Keywords: spinal cord stimulation; resting state functional magnetic resonance; voxel-based magnetic resonance morphometry
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- spinal cord stimulation (Experimental): The Vectris® SureScan® MRI lead will be connected to a RestoreSensor® SureScan® MRI neurostimulator.
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI

SUMMARY:
This study is an interventional prospective observatory single center trial, investigating the supraspinal effects of long term conventional SCS (60 Hz) and paresthesia-free high density SCS in failed back surgery syndrome (FBSS) patients with back and leg pain completed with resting state functional magnetic resonance (rs fMRI) and voxel-based magnetic resonance morphometry (VBM).

DETAILED DESCRIPTION:
When patient meets all inclusion criteria and no exclusion criteria, a neuroimaging protocol will be obtained at baseline, prior to trial implantation of SCS. At trial implantation a Vectris® SureScan® MRI 1x8 lead will be implanted, targeted by intraoperative mapping. This lead will be connected to a temporary extension cable and ENS.

Normal trial period will be respected based on the reimbursement rules in Belgium (4 weeks). When the patient is eligible for implantation of the definitive SCS system (more than 50% pain reduction and/or more than 50% reduction in pain medication), patient will undergo surgery for definitive implantation. Then the Vectris® SureScan® MRI lead will be connected to a RestoreSensor® SureScan® MRI neurostimulator.

After stabilisation of the stimulation parameters at least for more than 1 month, the second session of neuroimaging will occur (T1) with the RestoreSensor® SureScan® MRI neurostimulator in MRI mode. Minimal one month later ( 2 months after implantation of definitive SCS system) the patient will undergo the last session of neuroimaging (T2) with the stimulator in MRI mode. During that period prior to the MR-session, a new protocol will occur with paresthesia free high density SCS. The MRI protocol will occur after stabilisation of the stimulation parameters at least for more than 1 month. During the whole period, patients will fill in a VAS diary (back and leg pain separately) and at time of neuroimaging T1 and T2 a Likert-scale in order to evaluate the satisfaction grade of the patient. Additionally, patients will also wear during the whole period an Actiwatch, measuring sleep patterns and filling in questionnaires at B, T1 and T2 (Pittsburgh Sleep Quality Index (PSQI) and Holland Sleep Disorders Questionnaire (HSDQ).

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old.
* Subject is able and willing to comply with the follow-up schedule and protocol
* Diagnosis of FBSS with predominant leg pain (VAS) > 5) and non-dominant back pain.
* Cognitive and language functioning enabling coherent communication between the examiner and the subject;
* Failed conservative treatments for pain including but not limited to pharmacological therapy and physical therapy
* Stable neurologic function in the past 30 days
* In the opinion of the Investigator, the subject is psychologically appropriate for the implantation for an active implantable medical device
* Subject is able to provide written informed consent
* Subject speaks Dutch or French.

Exclusion Criteria:

* Female subject of childbearing potential is pregnant/nursing, or plans to become pregnant during the course of the trial
* Subject has had radiofrequency treatment of an intended target DRG within the past 3 months
* Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator, deep brain stimulator or intrathecal drug pump
* Subject is unable to operate the device or has no relative available.
* Subjects with indwelling devices that may pose an increased risk of infection
* Subject currently has an active infection
* Subject has, in the opinion of the Investigator, a medical comorbidity that contraindicates placement of an active medical device
* Subject has participated in another clinical investigation within 30 days
* Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
* Subject has been diagnosed with cancer in the past 2 years
* Life expectancy < 6 months
* Imaging (MRI, CT, x-ray) findings within the last 12 months that, in the Investigator's opinion, contraindicates lead placement
* Existing extreme fear for entering MRI
* General contraindication for MRI (pacemaker, etc…)
* Age male/female patient <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Grey Mater Volume assessed by Voxel-based morphometry analysis (based on MRI images) | The change between baseline and 1 month after definitive implantation (T1) and the change between baseline and 2 months after definitive implantation (T2).
Functional connectivity analysis using in-house developed software (based on MRI images) | The change between baseline and 1 month after definitive implantation (T1) and the change between baseline and 2 months after definitive implantation (T2).

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) pain diary | Three times every day (morning, afternoon and evening), starting 1 week before baseline measurements up to 2 months until study completion.
Objective sleep quality will be measured using the Actiwatch spectrum plus (Respironics). | The difference between 7 days at baseline before implantation and 7 days before T1 ( 1 month after definitive implantation) and 7 days before T2 ( 2 months after definitive implantation).
Subjective sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI) | The change between baseline and 1 month after definitive implantation (T1) and the change between baseline and 2 months after definitive implantation (T2).
Pain catastrophizing is assessed by the Pain Catastrophizing Scale (PCS) | The change between baseline and 1 month after definitive implantation (T1) and the change between baseline and 2 months after definitive implantation (T2).
Likert-scale in order to evaluate the satisfaction grade of the patient. | The change between baseline and 1 month after definitive implantation (T1) and the change between baseline and 2 months after definitive implantation (T2).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Vlaams Brabant, Belgium

REFERENCES:
- [Background] Rasche D, Siebert S, Stippich C, Kress B, Nennig E, Sartor K, Tronnier VM. [Spinal cord stimulation in Failed-Back-Surgery-Syndrome. Preliminary study for the evaluation of therapy by functional magnetic resonance imaging (fMRI)]. Schmerz. 2005 Nov;19(6):497-500, 502-5. doi: 10.1007/s00482-005-0388-9. German. PMID 15770488
- [Background] Stancak A, Kozak J, Vrba I, Tintera J, Vrana J, Polacek H, Stancak M. Functional magnetic resonance imaging of cerebral activation during spinal cord stimulation in failed back surgery syndrome patients. Eur J Pain. 2008 Feb;12(2):137-48. doi: 10.1016/j.ejpain.2007.03.003. Epub 2007 Oct 30. PMID 17977762
- [Background] Moens M, Sunaert S, Marien P, Brouns R, De Smedt A, Droogmans S, Van Schuerbeek P, Peeters R, Poelaert J, Nuttin B. Spinal cord stimulation modulates cerebral function: an fMRI study. Neuroradiology. 2012 Dec;54(12):1399-407. doi: 10.1007/s00234-012-1087-8. Epub 2012 Sep 2. PMID 22941431
- [Background] Moens M, Droogmans S, Spapen H, De Smedt A, Brouns R, Van Schuerbeek P, Luypaert R, Poelaert J, Nuttin B. Feasibility of cerebral magnetic resonance imaging in patients with externalised spinal cord stimulator. Clin Neurol Neurosurg. 2012 Feb;114(2):135-41. doi: 10.1016/j.clineuro.2011.09.013. Epub 2011 Oct 22. PMID 22018720
- [Background] Moens M, Marien P, Brouns R, Poelaert J, De Smedt A, Buyl R, Droogmans S, Van Schuerbeek P, Sunaert S, Nuttin B. Spinal cord stimulation modulates cerebral neurobiology: a proton magnetic resonance spectroscopy study. Neuroradiology. 2013 Aug;55(8):1039-1047. doi: 10.1007/s00234-013-1200-7. Epub 2013 May 12. PMID 23665999
- [Background] Qiu Y, Lv X, Su H, Jiang G, Li C, Tian J. Structural and functional brain alterations in end stage renal disease patients on routine hemodialysis: a voxel-based morphometry and resting state functional connectivity study. PLoS One. 2014 May 22;9(5):e98346. doi: 10.1371/journal.pone.0098346. eCollection 2014. PMID 24854737
- [Background] Chen Q, Yang W, Li W, Wei D, Li H, Lei Q, Zhang Q, Qiu J. Association of creative achievement with cognitive flexibility by a combined voxel-based morphometry and resting-state functional connectivity study. Neuroimage. 2014 Nov 15;102 Pt 2:474-83. doi: 10.1016/j.neuroimage.2014.08.008. Epub 2014 Aug 12. PMID 25123973
- [Background] Lui S, Deng W, Huang X, Jiang L, Ma X, Chen H, Zhang T, Li X, Li D, Zou L, Tang H, Zhou XJ, Mechelli A, Collier DA, Sweeney JA, Li T, Gong Q. Association of cerebral deficits with clinical symptoms in antipsychotic-naive first-episode schizophrenia: an optimized voxel-based morphometry and resting state functional connectivity study. Am J Psychiatry. 2009 Feb;166(2):196-205. doi: 10.1176/appi.ajp.2008.08020183. Epub 2008 Nov 3. PMID 18981063
- [Background] Becerra L, Sava S, Simons LE, Drosos AM, Sethna N, Berde C, Lebel AA, Borsook D. Intrinsic brain networks normalize with treatment in pediatric complex regional pain syndrome. Neuroimage Clin. 2014 Aug 10;6:347-69. doi: 10.1016/j.nicl.2014.07.012. eCollection 2014. PMID 25379449
- [Background] Yu R, Gollub RL, Spaeth R, Napadow V, Wasan A, Kong J. Disrupted functional connectivity of the periaqueductal gray in chronic low back pain. Neuroimage Clin. 2014 Aug 23;6:100-8. doi: 10.1016/j.nicl.2014.08.019. eCollection 2014. PMID 25379421